CLINICAL TRIAL: NCT03269942
Title: Results of Revascularization Versus Endovascular Flow Diversion in Treatment of Complex Intracranial Aneurysms of Anterior Circulation
Brief Title: Study of Complex Intracranial Aneurysm Treatment
Acronym: SCAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAT
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm; Flow Diverter; Cerebral Revascularization
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Cerebral Revascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Flow-Diversion (Active Comparator): Implantation of flow-diversion device
  Interventions: Procedure: Endovascular Flow-Diversion
- Cerebral Revascularization (Active Comparator): Cerebral revascularization procedure with trapping of aneurysm
  Interventions: Procedure: Cerebral Revascularization

INTERVENTIONS:
Procedure: Endovascular Flow-Diversion — Implantation of flow-diverter in treatment of complex aneurysms of anterior circulation.
  Arms: Endovascular Flow-Diversion
Procedure: Cerebral Revascularization — Cerebral revascularization with trapping of aneurysm in treatment of complex aneurysms of anterior circulation.
  Arms: Cerebral Revascularization

SUMMARY:
The investigator expects that endovascular flow-diversion is superior over revascularization by postoperative modified Rankin scale (mRS) in patients with complex intracranial aneurysms.

DETAILED DESCRIPTION:
Open, prospective, controlled randomized superiority trial is conducted. The hypothesis is that endovascular flow-diversion is better than revascularization in treatment of complex intracranial aneurysms by postoperative modified Rankin Scale (mRS). Sample size was measured by Fisher exact test. Depending on a type of the procedure, the patients are divided into two groups: Endovascular Flow Diversion Procedure (include 55 patients) and Revascularization Procedure (include 55 patients). Randomization is performed by random number generation.The study was approved by Institutional Review Board

ELIGIBILITY:
Inclusion Criteria:

* anterior circulation complex intracranial aneurysm
* neck is more than 4 mm wide
* dome/neck ratio of aneurysm equals or less than 2:1
* age less than 75 years
* ability to give informed consent (subject or legally authorized representative)
* aneurysm is suitable for treatment to both procedures

Exclusion Criteria:

* subarachnoid hemorrhage less than 30 days ago
* contraindications to endovascular treatment
* atypical aneurysms (mycotic, flow-related in patients with AVM, traumatic, false)
* informed consent refusal

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03-14 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
mRS | 6, 12 months after procedure
  Change from baseline modified Rankin Scale

SECONDARY OUTCOMES:
Complete aneurysm occlusion | 6, 12 months after procedure
  Measured as: complete occlusion or residual aneurysm (included neck remnant)
Major stroke (ischemic or hemorrhagic) or neurological death related to the treatment of the target aneurysm | 6, 12 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk Research Institution of Circulation Pathology, Novosibirsk, Russia